CLINICAL TRIAL: NCT06737263
Title: Comparison of BioHPP (High Performance Polymer) - vs Titanium- vs Zirconia Abutments A Randomized Controlled Clinical Trial
Brief Title: Comparison of BioHPP (High Performance Polymer) - vs Titanium- vs Zirconia Abutments
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BioHPP
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Peri-implant Soft Tissue Healing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BioHPP (Experimental): High Performance Polymer as abutment material
  Interventions: Device: BioHPP abutment
- Titanium (Active Comparator): Titanium as abutment material
  Interventions: Device: Titanium abutment
- Zirconia (Active Comparator): Zirconia as abutment material
  Interventions: Device: Zirconia abutment

INTERVENTIONS:
Device: BioHPP abutment — Patients in the test group receive abutments made of BioHPP
  Arms: BioHPP
Device: Titanium abutment — Patients in the control group receive abutments made of titanium
  Arms: Titanium
Device: Zirconia abutment — Patients in the control group receive abutments made of zirconia
  Arms: Zirconia

SUMMARY:
The project is a prospective, randomized, controlled study. The material BioHPP (High Performance Polymer) is compared with the gold-standard abutment materials titanium and zirconia in terms of peri-implant soft tissue healing.

DETAILED DESCRIPTION:
A total of 60 participants are divided into three groups of 20 persons each. One group receives BioHPP abutments, while the two control groups receive titanium or zirconia abutments.

The patients are provided with closed healing dental implants. After 3 months, following implant exposure and optical impression, the implants are restored with individual abutments.

Follow-up appointments are scheduled at 3, 6, 12, 24, and 36 months after implantation. During these visits, implant healing is assessed based on clinical parameters such as probing depth, plaque index, mean bone level, and bleeding on probing.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* The patients must be between 18 and 99 years old.
* non-smokers, former smokers, or light smokers (fewer than 10 cigarettes per day).
* ASA ( American Society of Anesthesiologists) Class I or II.
* There must be no pregnancy or breastfeeding period.
* the patients must have an edentulous section of up to 3 teeth in the maxillary or mandibular region, where it is possible to place an implant
* no allergy to any of the study-related materials

Exclusion Criteria:

* Patients under 18 or over 99 years old.
* Heavy smokers or former heavy smokers who quit less than five years ago
* Existing pregnancy or breastfeeding period.
* Individuals classified as ASA Class III to V.
* Presence of a polymer allergy.
* Patients with severe systemic diseases, immune deficiencies, or on corticosteroid medication.
* Patients undergoing local radiation or bisphosphonate therapy.
* Patients requiring sinus augmentation or soft tissue augmentation.
* Participation in another dental study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Mean Bone level | 36 months after implantation
  in millimeters

SECONDARY OUTCOMES:
Plaque index | 36 months after implantation
  in percent
Bleeding on probing | 36 months after implantation
  in percent
Probing depth | 36 months after implantation
  in millimeters
Occurrence of complications | 36 months after implantation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral Surgery and Radiology, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided